CLINICAL TRIAL: NCT01061229
Title: Homeopathic Drug Proving Trial
Acronym: HAMSV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ZS EK 15 - 287/09
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathic drug, potency C12 (Experimental)
  Interventions: Drug: Homeopathic drug C12
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Homeopathic drug C12 — Subjects in the intervention group are instructed to take five globules of the trial drug (potency C12), five times per day for a maximum of five days (5×5×5). The study medication is obtained from DHU (Germany), produced according to the Hahnemannian method. Subjects are asked to stop taking the medication, in agreement with their investigator, if they experience any of a predefined set of proving symptoms
  Arms: Homeopathic drug, potency C12
Other: Placebo — Placebo consists of pure sucrose globules (DHU, Germany) that are not potentiated nor impregnated with alcohol. The administration scheme is identical in the placebo control group to that of the intervention group.
  Arms: Placebo

SUMMARY:
The main aim of the study is to determine whether a homeopathic drug in the potency C12 provokes more characteristic homeopathic proving symptoms after three weeks compared to a placebo in healthy volunteers.

Secondary aims are to develop and to test a qualitative analysis methodology on which to base a definition for drug-specific (characteristic) symptoms and to compile a profile of characteristic homeopathic proving symptoms of the drug being trialled for therapeutic purposes.

This study protocol adapts the traditional homeopathic drug proving methodology to a modern clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors or medical students
* Not being treated for any acute or chronic diseases on the day of inclusion
* Written informed consent.

Exclusion Criteria:

* Pregnant women or nursing mothers
* Homeopathic treatment over the previous six weeks
* Participation in another clinical trial during the last six months
* Anyone with a personal or professional dependence on the study physician or sponsor
* Anyone who has been placed in hospital or other institution by authorities or decree

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome parameter is the number of characteristic proving symptoms per subject, derived from the qualitative data analysis of the homeopathic proving drug compared to placebo. | 3 weeks

SECONDARY OUTCOMES:
Total number of proving symptoms | 3 weeks
Number of serious adverse events | 3 weeks
Qualitative differences in the profiles of characteristic proving symptoms | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, Prof, MD, MBA, Principal Investigator — Charité University Berlin
Locations (1):
- Charité University, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Teut M, Hirschberg U, Luedtke R, Schnegg C, Dahler J, Albrecht H, Witt CM. Protocol for a phase 1 homeopathic drug proving trial. Trials. 2010 Jul 22;11:80. doi: 10.1186/1745-6215-11-80. PMID 20649979
- [Derived] Teut M, Dahler J, Hirschberg U, Luedtke R, Albrecht H, Witt CM. Homeopathic drug proving of Okoubaka aubrevillei: a randomised placebo-controlled trial. Trials. 2013 Apr 5;14:96. doi: 10.1186/1745-6215-14-96. PMID 23561008